CLINICAL TRIAL: NCT06996314
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation Combined With Slow-Paced Diaphragmatic Breathing on Postural Tachycardia Syndrome: A Randomized Controlled Trial
Brief Title: Effects of Auricular Vagus Nerve Stimulation Combined With Slow-paced Breathing on Individuals With Postural Orthostatic Tachycardia Syndrome.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Kapan (Other)
Responsible Party: Sponsor-Investigator, Ali Kapan, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1270/2024; KLP 2018025 (Other Grant/Funding Number: Austrian Science Fund)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS); Post-acute COVID-19 Syndromes
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TVNS + Slow-Paced Breathing (TVNS+SDB) (Active Comparator): Participants receive active transcutaneous auricular vagus nerve stimulation (taVNS) using electrodes placed at the cymba conchae, combined with guided slow-paced diaphragmatic breathing (0.1 Hz). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Interventions: Device: TVNS + Slow-Paced Breathing (TVNS+SDB)
- TVNS without Breathing Training (TVNS+NB) (Active Comparator): Participants receive active transcutaneous auricular vagus nerve stimulation (taVNS) using electrodes placed at the cymba conchae, combined with spontaneous breathing (no guided breathing exercises). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Interventions: Device: TVNS without Breathing Training (TVNS+NB)
- Sham TVNS + SDB (Active Comparator): Participants receive transcutaneous auricular vagus nerve stimulation using a sham protocol via electrodes placed at the cymba conchae, combined with guided slow-paced diaphragmatic breathing (0.1 Hz). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Interventions: Device: Sham TVNS + SDB
- Sham TVNS + NB (Sham Comparator): Participants receive transcutaneous auricular vagus nerve stimulation using a sham protocol via electrodes placed at the cymba conchae, combined with spontaneous breathing (no guided breathing exercises). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Interventions: Device: Sham TVNS + NB

INTERVENTIONS:
Device: TVNS + Slow-Paced Breathing (TVNS+SDB) — Participants receive active transcutaneous auricular vagus nerve stimulation (taVNS) using electrodes placed at the cymba conchae, combined with guided slow-paced diaphragmatic breathing (0.1 Hz). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Arms: TVNS + Slow-Paced Breathing (TVNS+SDB)
Device: TVNS without Breathing Training (TVNS+NB) — Participants receive active transcutaneous auricular vagus nerve stimulation (taVNS) using electrodes placed at the cymba conchae, combined with spontaneous breathing (no guided breathing exercises). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Arms: TVNS without Breathing Training (TVNS+NB)
Device: Sham TVNS + SDB — Participants receive transcutaneous auricular vagus nerve stimulation using a sham protocol via electrodes placed at the cymba conchae, combined with guided slow-paced diaphragmatic breathing (0.1 Hz). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Arms: Sham TVNS + SDB
Device: Sham TVNS + NB — Participants receive transcutaneous auricular vagus nerve stimulation using a sham protocol via electrodes placed at the cymba conchae, combined with spontaneous breathing (no guided breathing exercises). The intervention is performed daily at home for 12 weeks, with each session lasting 60 minutes.
  Arms: Sham TVNS + NB

SUMMARY:
This study investigates a non-pharmacological treatment approach for Postural Orthostatic Tachycardia Syndrome (POTS), a disorder of the autonomic nervous system characterized by an excessive increase in heart rate upon standing. POTS is commonly associated with symptoms such as dizziness, fatigue, cognitive difficulties, sleep disturbances, as well as anxiety and depression, which significantly impair quality of life.

This randomized, controlled clinical trial aims to evaluate whether combining transcutaneous auricular vagus nerve stimulation (taVNS) with slow-paced diaphragmatic breathing (at 0.1 Hz) provides greater therapeutic benefit compared to taVNS alone or sham stimulation.

A total of 100 participants will be recruited and randomly assigned to one of four groups (25 per group):

taVNS with slow-paced breathing,

taVNS with spontaneous (normal) breathing,

sham taVNS with slow-paced breathing, or

sham taVNS with spontaneous breathing.

Participants will perform the intervention daily at home for a duration of 12 weeks. Medical and psychological assessments will be conducted before and after the intervention, including measurements of heart rate, inflammatory cytokines, and patient-reported outcomes on sleep, mood, and quality of life.

The study is conducted at the Center for Public Health, Medical University of Vienna, and is open to individuals diagnosed with POTS, including those with coexisting Post-COVID-19 syndrome.

DETAILED DESCRIPTION:
Postural Orthostatic Tachycardia Syndrome (POTS) is a disorder of the autonomic nervous system characterized by an excessive increase in heart rate (≥30 bpm) within 10 minutes of standing, without a significant drop in blood pressure. Affected individuals frequently suffer from fatigue, dizziness, palpitations, cognitive dysfunction ("brain fog"), anxiety, depression, and sleep disturbances. These symptoms significantly impair daily functioning and quality of life.

Conventional pharmacological treatments often yield limited benefit and can lead to adverse effects, especially in individuals with complex autonomic dysregulation. Non-pharmacological approaches that target the autonomic nervous system more holistically and with fewer side effects are gaining increasing scientific interest.

This randomized, controlled clinical trial aims to investigate the effects of combining transcutaneous auricular vagus nerve stimulation (taVNS) with slow-paced diaphragmatic breathing at 0.1 Hz (six breaths per minute) as an integrative therapeutic strategy for individuals with POTS.

A total of 100 participants diagnosed with POTS will be randomly assigned (1:1:1:1) into four groups (25 per group):

taVNS combined with slow-paced diaphragmatic breathing (0.1 Hz)

taVNS combined with spontaneous breathing (no guided breathing exercises)

sham taVNS combined with slow-paced diaphragmatic breathing (0.1 Hz)

sham taVNS combined with spontaneous breathing (no guided breathing exercises)

All participants will undergo standardized instruction in the use of the stimulation device and, where applicable, in breathing technique by a trained therapist. The intervention will be performed daily at home for 12 weeks. taVNS is administered for 60 minutes per session using a CE-certified medical device (Nurosym™), with stimulation parameters set at 20 Hz and 200 µs pulse width. For those in the breathing groups, the slow-paced breathing is guided via a mobile app and performed for 10 minutes in the first 4 weeks and 15 minutes in the final weeks.

To evaluate the intervention's effects, a comprehensive set of physiological and psychological parameters will be assessed before and after the 12-week intervention period, including:

Change in heart rate response to orthostatic challenge (Tilt Test)

Capnography (end-tidal CO₂ monitoring) during the Tilt Test to assess ventilatory compensation and respiratory dysregulation

Cerebral tissue oxygenation measured by near-infrared spectroscopy (NIRS) during orthostatic testing to evaluate cerebral perfusion

Heart rate variability (HRV)

Serum levels of inflammatory cytokines (TNF-α, IL-6, IL-8, CRP)

Self-reported symptom burden (Malmö POTS Symptom Score)

Sleep quality (PSQI)

Health-related quality of life (SF-36)

Psychological distress (DASS-21)

Daily activity and resting heart rate (7-day wearable device)

Handgrip strength as a marker of physical capacity

Participants will also be monitored for adherence and potential adverse events. The sham taVNS groups will use identical devices delivering subthreshold stimulation to maintain blinding.

The study is conducted at the Center for Public Health, Medical University of Vienna. Eligible participants must have a confirmed diagnosis of POTS, with or without post-COVID syndrome, and meet the study's inclusion criteria. Randomization is stratified by sex and post-COVID status to ensure balance across treatment arms.

This trial aims to determine whether the integrative approach of vagal stimulation and paced breathing can enhance autonomic regulation, improve cerebral perfusion, reduce inflammation, and improve psychological outcomes in individuals with POTS. The results may offer an evidence-based foundation for non-invasive neuromodulation in the management of autonomic disorders.

ELIGIBILITY:
Inclusion Criteria:

Formal diagnosis of Postural Orthostatic Tachycardia Syndrome (POTS), confirmed by clinical criteria: a sustained increase in heart rate (HR) of ≥30 bpm within 10 minutes of standing, without orthostatic hypotension.

History of POTS diagnosis for at least 6 months.

Participants with Post-acute COVID-19 syndrome may be included if they meet the formal POTS criteria. These participants will be stratified based on the presence or absence of Post-Exertional Malaise (PEM).

Stable medication for POTS (same dosage/class) for at least 4 weeks before enrollment.

Willingness and ability to provide informed consent.

Screening of Undiagnosed Participants:

Suspected POTS based on clinical symptoms (e.g., dizziness, fatigue, syncope, brain fog, palpitations, exercise intolerance) persisting ≥6 months.

Preliminary Schellong test by study team.

If criteria are met, referral to a specialist (neurology or cardiology) for diagnostic confirmation.

Inclusion only after specialist-confirmed POTS diagnosis.

Exclusion Criteria:

Significant hypertension (BP >150/100 mmHg supine or standing).

Orthostatic hypotension: drop in BP >20 mmHg systolic or >10 mmHg diastolic upon standing.

Recent stroke or myocardial infarction (within 6 months).

Significant immunological or hematological disorders.

Severe anemia (hematocrit <28%).

History of vagotomy.

Pregnancy or lactation.

Inability or unwillingness to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate From Supine to Standing (Delta HR) After 12 Weeks of Daily taVNS With or Without Slow-Paced Breathing in Individuals With POTS | Change in Heart Rate (Delta HR) from Supine to Standing at Baseline and Week 12
  Heart rate (HR) is continuously recorded via 12-lead ECG during a standardized Tilt test. Participants lie supine for 25 minutes and then stand upright for 10 minutes. The average HR from the last 10 minutes supine and the 10-minute standing phase is calculated. The primary outcome, Delta HR, is defined as the difference between upright and supine HR. This measure reflects autonomic cardiovascular response and is assessed before and after the 12-week intervention phase.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kapan, PhD, Principal Investigator — Medical University of Vienna, Center for Public Health,

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. According to the informed consent and data protection requirements, data may only be used within the study and by authorized parties. No data will be shared outside the study team or transferred to third parties, including for secondary analysis or outside the EU.

REFERENCES:
- See also: Related Info — https://www.meduniwien.ac.at/web/